CLINICAL TRIAL: NCT01530256
Title: An Exploratory Phase 1/2 Clinical Trial Evaluating ALD518 in Subjects With Glucocorticoid-Refractory Acute Graft vs. Host Disease (GVHD) After Allogeneic Hematopoietic Stem Cell Transplant (HSCT)
Brief Title: Exploratory Safety Study of ALD518 in Subjects With Steroid-refractory Acute Graft Versus Host Disease (GVHD)
Acronym: ALD518-010
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The trial was terminated in line with the endpoint committee charter.
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALD518-CLIN-010
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Acute GvHD
Keywords: allograph; steroid refractory
MeSH Terms: interventions — clazakizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALD518 (Experimental)
  Interventions: Biological: ALD518

INTERVENTIONS:
Biological: ALD518 — 160 mg IV q 4 weeks for 4 doses
Biological: ALD518 — 320 mg IV q 4 weeks for 4 doses
Biological: ALD518 — 640 mg IV q 4 weeks for 2 doses

SUMMARY:
The purpose of this study is to determine the safe and tolerable, biologically active, and potentially effective doses(s) of ALD518 in subjects with acute GVHD, who have failed to respond to glucocorticosteroids, for further investigation in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Glucocorticosteroid refractory acute GVHD Grade 2-4
* Prior corticosteroid therapy at > 1.0mg/kg methylprednisolone or equivalent for minimum of 3 and maximum of 14 days
* Karnofsky Performance Satus Scale ≥ 50%
* Adequate laboratory testing at screening

Exclusion Criteria:

* Subjects having Stage 1 skin acute GVHD
* Subjects with Stage 3 or 4 liver GVHD
* Prior EBV associated malignancy
* Prior or current Hepatitis B or C
* Prior or active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier San Martin, MD FRCP, Study Director — Alder Biopharmaceuticals, Inc.
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Loyola Medical Center, Maywood, Illinois
  - Washington University, St Louis, Missouri
  - The Ohio State University, Columbus, Ohio
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial was terminated after only 3 participants received the 160 mg dose.
Groups:
- ALD518: ALD518: 160 mg intravenous (IV) once every (q) 4 weeks for 4 doses
Period: Overall Study
Arm/Group | ALD518
Started | 3
Completed | 1
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | ALD518
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Including Infections and Loss of Engraftment
Time Frame: Through Week 24
Measure: Number; unit: participants
Arm/Group | ALD518
Number analyzed (Participants) | 3
participants | 3

2. Primary Outcome: Number of Participants With Acute GVHD Response at Week 4
Description: Includes calculation of both complete and partial response. Complete response = functional grade of 0 for the GVHD grading in all evaluable organs. Partial response = improvement by one or more functional grades in one or more organs involved with GVHD symptoms without progression in others, or a very good partial response which is a partial response plus all of the following: (1) skin - active erythematous rash involving less than 25% of body surface, (2) liver - total bilirubin <2 mg/dL or a 25% reduction from baseline (if >2 mg/dL), (3) gut - greater than or equal to 75% reduction in daily stool volume.
Time Frame: Week 4
Population: 2 of 3 participants died before Week 4 so could not be assessed
Measure: Number; unit: participants
Arm/Group | ALD518
Number analyzed (Participants) | 1
participants | 0

3. Secondary Outcome: Number of Participants With Relapse of Underlying Malignant Disease
Time Frame: Through Week 24
Measure: Number; unit: participants
Arm/Group | ALD518
Number analyzed (Participants) | 3
participants | 0

4. Secondary Outcome: Number of Participants With Overall Survival
Time Frame: Through Week 24
Measure: Number; unit: participants
Arm/Group | ALD518
Number analyzed (Participants) | 3
participants | 1

5. Secondary Outcome: Change in Patient Reported Outcomes as Measured by the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) Questionnaire Score
Description: The FACT-BMT assesses bone marrow transplant related concerns. The total score is the sum of sub-scale scores for 5 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, and Bone Marrow Transplantation Subscale. Within each domain, a 5-point Likert-type scale (from 0-4) is used to measure the responses for each question. After taking into account reverse scores for questions constructed in a negative form, the subscale score for each domain is calculated by multiplying the sum of the item scores by the number of items in the subscale, then dividing by the number of items answered. The final score for FACT-BMT ranges from 0 to 148. Higher scores indicate better quality of life.
Time Frame: Up to 20 weeks
Measure: Number; unit: score on a scale
Arm/Group | ALD518
Number analyzed (Participants) | 2
score on a scale
  Participant 1 (Day 0) | 93
  Participant 1 (Week 4) | 96
  Participant 1 (Week 12) | 102
  Participant 1 (Week 20) | 113
  Participant 2 (Day 0) | 55

ADVERSE EVENTS:
Time Frame: Up to death or termination of study (approximately 139 days).
Arm/Group | ALD518
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALD518 (N=3)
Renal failure acute (Renal and urinary disorders) | 2 (3)
Sepsis (Infections and infestations) | 1 (2)
Retinal detachment (Eye disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALD518 (N=3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
International normalized ratio increased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Oedema peripheral (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Formal analyses were not conducted. Profiles of each enrolled subject were produced. Due to a limited number of samples, pharmacokinetics and anti-ALD518 antibodies analyses were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No